CLINICAL TRIAL: NCT03316430
Title: Prospective Study : Podocyturia as Predictive Factor for Pre-eclampsia
Brief Title: Podocyturia as Predictive Factor for Pre-eclampsia
Acronym: PEPOD1
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0516
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients coming before 16 weeks of gestation at their first planned prenatal visit at the Hôpital Femme Mère Enfant, who planned to deliver at the Hôpital Femme Mère Enfant
  Interventions: Other: Podocyturia quantification

INTERVENTIONS:
Other: Podocyturia quantification — Podocyturia quantification at first planned prenatal care visit before 16 weeks of gestation

SUMMARY:
Pre-eclampsia is an hypertensive disorder appearing during pregnancy, inducing serious maternal, fetal and neonatal mortality and morbidity. Podocyn could be identified in the urine, before proteinuria, a key element in the diagnostic of pre-eclampsia. Preventive treatment using aspirin could be administrated in early pregnancy. We hypothesized that podocyturia could be an early indicator of preeclampsia. This is a prospective, non-interventional, monocentric study.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years or more
* single pregnancy
* first planned prenatal visit before 16 weeks of gestation
* planned delivery at Hôpital Femme Mère Enfant in Lyon, France
* patient receiving information and non opposition to participate

Exclusion Criteria:

* multiple pregnancy
* pregnancy stopped
* antecedent of nephropathy
* inability to understand information provided
* prisoner or under administrative supervision
* fetal malformation, chromosomal anomalies
* preterm delivery for other reason that any hypertensive disorder of pregnancy or Intrauterine growth restriction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients coming before 16 weeks of gestation at their first planned prenatal visit at the Hôpital Femme Mère Enfant, who planned to deliver at the Hôpital Femme Mère Enfant
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of pre-eclampsia | At childbirth (around 8 months)
  Occurrence of pre-eclampsia during pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of obstetrics, Femme Mère Enfant Hospital, Lyon, France, Bron, France

IPD SHARING:
Plan to Share IPD: No